CLINICAL TRIAL: NCT04918095
Title: CareCOPD - Chronic Obstructive Pulmonary Disease (COPD) Home Monitoring for Early Exacerbation Detection
Brief Title: CareCOPD - COPD Home Monitoring Study
Status: Recruiting | Type: Observational
Sponsor: Cognita Labs LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CareCOPD20
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Moderate-Severe COPD: COPD patients diagnosed GOLD 2- 3, C- D for moderate-severe, poorly controlled
  Interventions: Device: CareCOPD Platform

INTERVENTIONS:
Device: CareCOPD Platform — The subjects will be provided with CareCOPD devices for home monitoring of airway impedance, medication use, and symptoms data.

SUMMARY:
This is a pilot study to demonstrate early validation of objective home-monitoring of Chronic obstructive pulmonary disease (COPD) patients by combining accurate and relevant patient data of medication and lung function (lung impedance) through patient-facing devices.

DETAILED DESCRIPTION:
The study goals are to demonstrate early validation of objective home-monitoring of COPD patients using CareCOPD mature devices, paving way for follow-up work of care integration and larger studies. The data will consist of time-series airway obstruction parameters, medication quality, and symptoms data to detect correlations with exacerbation events. 50 COPD patients (diagnosed GOLD 2- 3, C- D for moderate-severe, poorly controlled) will be monitored for 6 months. A successful outcome will be improved acute exacerbation of COPD or AECOPD detection of at least one day earlier than patient-reported assessment (COPD Assessment Test or CAT, modified Medical Research Council or mMRC questionnaires) and false positives of <20%.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following criteria are eligible for enrollment as study participants:

* Males and females over the age of 40 years.
* physician-diagnosed COPD classified as GOLD 2-3, C-D for at least 1 year.
* Using rescue medications at home delivered by a metered-dose inhaler or MDI.
* Speak, read, and understand English.
* Able to understand study requirements and comply with study procedures.
* Ability to operate a smartphone or tablet (for questionnaire and symptoms input).

Exclusion Criteria:

Subjects who meet any of these criteria are not eligible for enrollment as study participants:

* Physically disabled such that they are incapable of performing forced oscillometry test (for airway impedance measurement)
* Physically disabled such that they are incapable of using metered-dose inhalers.
* Suffer from any visual, hearing, or cognitive impairment that cannot be corrected enough to operate the CareCOPD devices properly. Mild/moderate vision loss and mild hearing loss may be included with appropriate corrective measures that do not affect the device usage.
* Suffering from serious uncontrolled medical conditions that may interfere with study conduct.
* Continuous home Oxygen use for greater than 16 hours/day.
* Inability or unwillingness of the participant to give written informed consent.
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD primarily affects and has adverse events for adults over the age of 40 based on prior COPD literature. Further, this study is observational, to study correlations between CareCOPD platform collected data and AECOPD. AECOPD is more frequent in older adults and will provide more data for the limited pilot study. Therefore, subjects in the study will exclusively be 40 years of age and older. There is no upper limit on age. As the pilot study expands to include interventions from the CareCOPD platform, the age range may be modified to include all subjects having COPD.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-11-09 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of AECOPD | 6 months
  Percentage of AECOPDs detected by CareCOPD platform

SECONDARY OUTCOMES:
Average number of days before AECOPD detection | 6 months
False positivity rate | 6 months
  False positivity rate in the detection of AECOPD

CONTACTS AND LOCATIONS:
Locations (1):
- Ventura County Medical Center, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: No